CLINICAL TRIAL: NCT00844818
Title: Using the Postpartum Hospital Stay to Address Mother's and Father's Smoking: the NEWS Study
Brief Title: An Intervention to Address Parental Smoking During the Postpartum Hospitalization.
Acronym: NEWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Jonathan Winickoff, MD, MPH, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004P002104
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Tobacco Use; Parental Smoking
Keywords: smoking cessation; parents
MeSH Terms: conditions — Tobacco Use; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Moms and dads who were current smokers (1 cigarette, even a puff, in past 30 days) or recent quitters (smoked since one month prior to conception)
- Intervention Group (Experimental): Moms and dads who were current smokers (1 cigarette, even a puff, in past 30 days) or recent quitters (smoked since one month prior to conception)
  Interventions: Behavioral: Telephone Quitline Enrollment

INTERVENTIONS:
Behavioral: Telephone Quitline Enrollment — The intervention included a brief motivational interview (MI), enrollment in the proactive state quitline, and follow-up faxes to the pediatric, OB, and PCP providers with tailored treatment messages.
  Arms: Intervention Group

SUMMARY:
The purpose of the study is to find better ways to help parents quit smoking, thus improving their own health, the health of their children, and the health of other family members. This study tested the feasibility and acceptability of enrolling parents into a telephone quitline during postpartum hospitalization. Half of the parents in the study received quit smoking assistance (intervention group), and half of the parents did not (control group). The percentage of parental smokers who are enrolled in quit smoking programs by the study follow-up will be greater in the intervention group than in the control group.

DETAILED DESCRIPTION:
This is a randomized control trial to test the feasibility and efficacy of modifying hospital staff practices on the postpartum floor and intervening with parents before hospital discharge to help them quit smoking. Over 14 months, we assessed the smoking status of both parents of all newborns delivered at 1 hospital. Moms and dads who were current smokers (1 cigarette, even a puff, in past 30 days) or recent quitters (smoked since one month prior to conception) were eligible for the study. Enrolled parents were randomly assigned to the control or intervention group. The intervention included a brief motivational interview (MI), enrollment in the proactive state quitline, and follow-up faxes to the pediatric, OB, and PCP providers with tailored treatment messages.

ELIGIBILITY:
Inclusion Criteria:

* Parents of newborns delivered at MGH ("parent" includes the mother, father or another legal guardian) who are: a) current smokers (have smoked, even a puff, within the last 30 days and/or b) recent quitters (have smoked, even a puff, since 30 days prior to conception);
* Telephone access;
* English competency, adequate to participate in the interview;
* Massachusetts resident for next 3 months (from date of consent).

Exclusion Criteria:

* Non-smokers or parents who have not smoked since before one month prior to conception (cessation great than 10 months);
* Non-English speaking;
* Non-Massachusetts residents;
* Any family with critically ill mother or infant that the obstetrical nurse practitioner does not feel is appropriate to be approached;
* Decline participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2005-02; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Winickoff, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States